CLINICAL TRIAL: NCT07028450
Title: Effects of Proactive Calls: A Randomized Controlled Study
Brief Title: Effects of Proactive Call to Customers of Norsk Rikstoto (Horse Gambling Operator in Norway): A Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Norsk Rikstoto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Spillforsk25/1
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Gambling Problem
Keywords: Gambling Problem; Proactive calls; Randomized controlled trial; mini-intervention

STUDY DESIGN:
Intervention Model Description: The two arms/conditions involves one proactive phone call or a control condition
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One proactive call (Experimental): The call is based on principles of motivating interviewing and will in addition encourage the recipient to change his/hers gambling behavior (e.g., lower pre-set loss limits).
  Interventions: Behavioral: Proactive call
- Control (No Intervention): No contact/not reaching out

INTERVENTIONS:
Behavioral: Proactive call — The proactive call will be based on the principles of motivational interviewing. The content of the call comprises: 1) Asking the gambler/recipient to reflect on their gambling behavior, 2) providing to the gambler/recipient an overview of their gambling account and financial history, 3) offering to the gambler/recipient information about responsible gambling tools, such as setting lower limits, locking limits, taking a break, or self-exclusion, and 4) providing to the gambler/recipient information about relevant support services and the Gamban tool in cases where a need is expressed.
  Arms: One proactive call

SUMMARY:
Customers/gamblers gambling at Norsk Rikstoto (gambling monopolist in Norway providing horse gambling products with potential gambling problems will be randomly allocated to receive a proactive phone call (encouraging them to change their gambling behavior - e.g., be lowering the loss limit) or to a control condition. Outcomes will be short and long terms registered gambling behavior.

DETAILED DESCRIPTION:
Norsk Rikstoto (gambling monopolist in Norway providing horse gambling products) enforces registered play, hence all gambling transactions and outcomes of stakes of all customers are registered and stored for 5 years. Based on daily algorithms high risk gamblers are identified. Gamblers 18-35 years who for at least 5 of the last 30 days have been identified as high risk gamblers will according to a 1.5:1 ratio be allocated to a proactive call condition or to a control condition.

The call will be based on principles from motivating interviewing and will contain encouragements to alter gambling behavior (e.g., lowering loss limits). Primary outcome comprises theoretical loss (total bet x house advantage ((100% - payback%) / 100)). Secondary outcomes comprises total stakes made by the customer and loss percentage (proportion of stake that is lost). Baseline data comprises gambling behavior the 30 days before the call. Short-term effects comprise cumulative registered gambling behavior the first 90 days after the call whereas long-term effects consist of cumulative registered gambling behavior day 91-180 after the call. A random block design will be used where 15 eligible customers each week will be allocated either to the proactive call condition (n=9) or to the control condition (n=6).

ELIGIBILITY:
Inclusion Criteria:

* Being identified (based on an algorithm used by Norsk Rikstoto/the gambling provider) as a high risk gambler at least 5 of the last 30 days

Exclusion Criteria:

* None

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Theoretical loss | Change from baseline (30 days before the call) to day 1-90 after the call (short-term effect) and change from baseline (30 days before the call) to day 91-180 after the call (long-term effect).
  Total bet x house advantage ((100%-payback%) / 100)

SECONDARY OUTCOMES:
Total stake | Change from baseline (30 days before the call) to the first 90 days after the call (short term) and change from baseline to day 91-180 after the call
  Total amount of money staked
Loss percentage | Change from baseline (30 days before the call) to day 1-90 after the call (short-term effect) and change from baseline (30 days before the call) to day 91-180 after the call (long-term effect).
  Percentage of stakes that are lost

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Department of Psychosocial Science, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Researchers may contact the principle investigator and ask for access to the data in anonymous form
Supporting Information: Study Protocol, SAP